CLINICAL TRIAL: NCT01400204
Title: A Naturalistic Study Comparing the Hangover Effects of MDMA, Other Drugs, and Alcohol in a Sample of Recreational Polydrug Users
Brief Title: Naturalistic Study Into the Hangover Effects of MDMA
Status: Completed | Type: Observational
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Responsible Party: Joris C Verster, PhD, Utrecht University
Other Study IDs: ppo-010-212
Record Dates: First submitted 2011-07-21; First posted 2011-07-22 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Hangover
Keywords: hangover; next day effects; MDMA; Alcohol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MDMA: poly drug users that used MDMA at New Years Eve
- Other Drugs: poly drug users that used drugs at New Years Eve, but not MDMA
- Alcohol: poly drug users that used no drugs at New Years Eve, but did consume alcohol

SUMMARY:
The aim of the study is to compare hangover effects of MDMA users versus those who used other drugs, or alcohol only at New Year's Eve. The week after New Years Eve, every day participants complete a questionnaire about the presence and severity of potential hangover symptoms. At day 1, demographics and alcohol and drug use at New Years Eve were recorded. On day 7, the Brief Symptom Inventory (BSI) is completed to asses last weeks mood. After 4 weeks, after a drug-free week, the BSI is completed again to serve as a reference.

DETAILED DESCRIPTION:
A convenience sample was invited by e-mail to participate in the study, via the organizer of a private New Years Party.It was attempted to include as much participants as possible. Hence, no sampling method was applied when recruiting participants.

ELIGIBILITY:
Inclusion Criteria:

* poly drug user
* 18+ years old

Exclusion Criteria:

* mental or physical illness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recreational poly-drug users who were guests at a privat New Years Eve party
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2010-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joris C Verster, PhD, Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Utrecht, Netherlands